CLINICAL TRIAL: NCT07230236
Title: Investigation of the Relationship Between LS Chirp ABR and Comprehension In Noise Skills In Individuals With Suspected Hidden Hearing Loss
Brief Title: Relationship Between LS Chirp ABR and Speech-in-Noise Skills in Hidden Hearing Loss
Status: Recruiting | Type: Observational
Sponsor: Istanbul University - Cerrahpasa (Other)
Collaborators: Medipol University (Other)
Responsible Party: Principal Investigator, Cem Yeral, Research Assistant Cem Yeral, Istanbul University - Cerrahpasa
Other Study IDs: 2025/379
Record Dates: First submitted 2025-10-02; First posted 2025-11-17 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-11

CONDITIONS: Hidden Hearing Loss; Cochlear Synaptopathy
Keywords: hidden hearing loss; cochlear synaptopathy; Level-Specific (LS) Chirp ABR; Hearing In Noise Test (HINT)
MeSH Terms: conditions — Hearing Loss, Hidden

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 10 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Control group: Inclusion Criteria
  Being between 20 and 60 years of age, Having bilateral pure-tone audiometry averages (500-1000-2000-4000 Hz) within the normal range (≤25 dB HL), Having no tinnitus or auditory complaints, Scoring 21 or above on the MoCA test, Having no emotional or neurological problems that could interfere with the tests.
  Exclusion Criteria
  Presence of peripheral and/or central hearing loss, Presence of somatosensory tinnitus, Presence of emotional and/or neurological problems that could interfere with the tests.
- First study group: Inclusion Criteria
  Being between 20 and 60 years of age, Having bilateral pure-tone audiometry averages (500-1000-2000-4000 Hz) within the normal range (≤25 dB HL), Having a chronic tinnitus complaint (≥3 months), Scoring 21 or above on the MoCA test, Having no emotional or neurological problems that could interfere with the tests.
  Exclusion Criteria
  Presence of peripheral and/or central hearing loss, Presence of somatosensory tinnitus, Presence of emotional and/or neurological problems that could interfere with the tests.
- Second study group: Inclusion Criteria
  Being between 20 and 60 years of age, Having bilateral pure-tone audiometry averages (500-1000-2000-4000 Hz) within the normal range (≤25 dB HL), Having no chronic tinnitus complaint, The mean scores on the questions assessing the ability to understand speech in noise in the "Speech Perception" subscale of the SSQ (Speech, Spatial, and Hearing Quality Scale) are below the normative value, Scoring 21 or above on the MoCA test, Having no emotional or neurological problems that could interfere with the tests.
  Exclusion Criteria
  Presence of peripheral and/or central hearing loss, Presence of somatosensory tinnitus, Presence of emotional and/or neurological problems that could interfere with the tests.

SUMMARY:
It is known that the underlying problem in Hidden Hearing Loss (HHL) is cochlear synaptopathy (CS) and that low-spontaneous-rate auditory nerve fibers play an important role in this pathology. Therefore, it is suggested that low-spontaneous-rate auditory nerve fibers are damaged in HHL. Consequently, LS CE-Chirp-evoked ABR and HINT, which assesses CS by presenting stimuli of varying intensities and characteristics to provide information about auditory nerve fibers, will be used to evaluate participants both objectively and subjectively.

Aim of the study:

The main aim of this study is to investigate the relationship between the amplitude and latency values obtained with LS CE-Chirp-stimulated ABR and the critical Signal-to-Noise Ratio (SNR) obtained from the Hearing in Noise Test (HINT) in individuals suspected of having HHL.

Hypotheses

H0: In individuals suspected of having HHL, there is no relationship between the amplitude values of waves I, III, and V obtained with LS CE-Chirp ABR at 80, 90, and 100 dBnHL and the I/V amplitude ratio and the critical SNR obtained from HINT.

H1: In individuals suspected of having HHL, there is a relationship between the amplitude values of waves I, III, and V obtained with LS CE-Chirp ABR at 80, 90, and 100 dBnHL and the I/V amplitude ratio, and the critical SNR obtained from HINT.

Expected Results:

The study will reveal how LS CE-Chirp stimulation affects ABR results in individuals suspected of having HHL, and the relationship between these results and HINT results will be examined. In this way, HHL will be evaluated both objectively (LS CE-Chirp ABR) and subjectively (HINT). Based on the findings, scientific outputs such as publications or projects are targeted.

Importance:

HHL has recently attracted increasing attention as a condition that significantly affects daily life. In today's world, where noise and noisy environments are prevalent, disadvantages arise in many aspects, particularly in communication. Therefore, the findings obtained in this study may contribute to a better understanding of HHL.

DETAILED DESCRIPTION:
Hidden Hearing Loss (HHL) is defined as the presence of normal pure-tone audiometric thresholds accompanied by self-reported listening difficulties, most notably problems understanding speech in noisy environments. Recent neurophysiological and histopathological evidence suggests that this condition is associated with cochlear synaptopathy-selective loss or dysfunction of the synapses between inner hair cells and low-spontaneous-rate (low-SR) type I auditory nerve fibers. Low-SR fibers are crucial for encoding suprathreshold acoustic signals and preserving speech perception in noise. Damage to these fibers can occur from noise exposure, aging, or other metabolic factors even when outer hair cells remain intact, thereby leaving conventional audiometry within normal limits.

Auditory Brainstem Response (ABR) testing provides an objective measure of neural synchrony along the auditory pathway. The amplitude and latency of early ABR waves, particularly Waves I, III, and V, reflect the temporal integrity of auditory nerve and brainstem transmission. Among these, Wave I amplitude is considered a peripheral marker of auditory nerve fiber activity, while Wave V represents the summated output of higher brainstem nuclei. A reduction in Wave I amplitude with preserved Wave V amplitude, or a decreased I/V ratio, is interpreted as an electrophysiological signature of cochlear synaptopathy.

Traditional ABR using click stimuli synchronizes neural responses primarily from the basal cochlear region. The introduction of chirp stimuli aimed to improve neural synchrony by compensating for cochlear travel-time delays. The Level-Specific (LS) CE-Chirp stimulus designed by Claus Elberling and Don allows the amplitude of Wave V to remain robust across intensities while providing frequency-specific timing. Yet, at high levels (80-100 dB nHL), LS CE-Chirp responses may demonstrate altered growth functions and latency patterns, potentially revealing subtle differences in suprathreshold neural coding compared to conventional clicks.

The current study adopts an observational, cross-sectional, correlational design to investigate whether electrophysiological indices derived from LS CE-Chirp-stimulated ABR are associated with behavioral speech-in-noise performance in individuals suspected of HHL. Participants with normal pure-tone thresholds will undergo both ABR and the Hearing In Noise Test (HINT), enabling exploration of the relationship between amplitude and latency measures of ABR waves and the critical signal-to-noise ratio (SNR-50) obtained behaviorally.

The scientific rationale for the study stems from the premise that reduced neural output from low-SR auditory fibers manifests as smaller Wave I amplitudes at high stimulation levels, producing diminished I/V ratios and flattened amplitude-growth slopes. These physiological patterns are expected to parallel poorer speech-in-noise perception, reflected by elevated SNR-50 values on HINT. Demonstrating a significant correlation between ABR parameters and HINT outcomes would thus support the hypothesis that LS CE-Chirp ABR can serve as an objective marker of suprathreshold auditory coding deficits in HHL.

Participants will be recruited from audiology clinics and university hearing research laboratories. Three subgroups will be studied:

1. A control group with normal hearing and no tinnitus or listening complaints;
2. A tinnitus group with chronic subjective tinnitus (≥ 3 months) but normal hearing thresholds; and
3. A speech-in-noise complaint group reporting difficulty understanding speech in background noise despite normal thresholds and no tinnitus.

Eligibility criteria include ages 20-60 years, bilateral air-conduction thresholds ≤ 25 dB HL at 0.5-4 kHz, normal immittance results, and MoCA ≥ 21. Individuals with peripheral or central hearing loss, somatosensory tinnitus, neurological disorders, or significant emotional/psychiatric conditions will be excluded. Approximately 63 participants (21 per group) are planned, as determined by G*Power analysis (effect size 0.5, α = 0.05, power = 0.80). Recruitment status is active.

All participants will provide written informed consent. Testing will occur in a sound-attenuated booth. The assessment sequence includes:

Montreal Cognitive Assessment (MoCA) for cognitive screening;

Speech, Spatial and Qualities of Hearing Scale (SSQ) or its Turkish adaptation for subjective speech-perception profiling;

Pure-tone audiometry to confirm normal thresholds;

Threshold Equalizing Noise (TEN) test to screen for cochlear dead regions (control measure, not analyzed);

Immittance and acoustic reflexes to confirm middle-ear integrity;

LS CE-Chirp and Click ABR recordings; and

HINT administration in free-field conditions.

ABR recordings will be obtained monaurally using the Neurosoft Neuro-MEP-4 system. Disposable surface electrodes will be applied after skin preparation with Nuprep gel: active (Cz or Fz), reference (ipsilateral mastoid A1/A2 or earlobe), and ground (FPz or AFz). Electrode impedance will be maintained below 3 kΩ and balanced across channels. Insert earphones will deliver alternating-polarity stimuli to minimize cochlear microphonic artifacts.

For both Click and LS CE-Chirp stimuli, recordings will be made at 80, 90, and 100 dB nHL using a 21.1 stimuli/s repetition rate; additional short blocks may use 11.1 or 61.1 /s to examine neural adaptation. The recording filter will be 100-3000 Hz (12 dB/octave), artifact rejection ± 35-40 µV, and analysis window 0-15 ms (pre-stimulus -2 ms). Each condition will comprise 2000-4000 sweeps averaged twice for replicability; recordings with residual noise > 20 nV rms or inter-replicate discrepancy > 15 % will be repeated. Insert-earphone tubing delay (≈ 0.9 ms) will be compensated in latency calculations.

Wave peaks I, III, and V will be identified independently by two blinded examiners. Amplitude and latency measures will be extracted for each wave at each intensity, and V/I amplitude ratios will be computed. LS CE-Chirp responses are expected to show larger Wave V amplitudes at lower intensities and potential amplitude saturation at higher intensities, providing a basis for evaluating suprathreshold neural synchronization.

The HINT will consist of 25 sentence lists (10 sentences each, total 250 sentences). Speech will be presented at variable levels while background noise is held constant at 65 dB SPL. The adaptive algorithm adjusts sentence level according to participant accuracy, converging on the critical SNR (dB) where 50 % of sentences are correctly repeated. Testing will be conducted with the participant seated 1 meter from the loudspeaker at 0° azimuth in a calibrated free-field environment.

Data from ABR and HINT will be linked for correlational analysis. For each participant, "better-ear" ABR metrics (based on higher Wave I amplitude) will be paired with binaural HINT performance to reflect real-world auditory integration.

Data Analysis Plan

Data will be analyzed using the Statistical Package for the Social Sciences (SPSS v27). The normality of variable distributions will be verified using the Kolmogorov-Smirnov test. Depending on the results, parametric or non-parametric statistics will be applied. For group comparisons, one-way analysis of variance (ANOVA) will be used for normally distributed variables, and the Kruskal-Wallis test will be applied for non-normal distributions. When significant effects are found, appropriate post-hoc pairwise comparisons with Bonferroni or Dunn corrections will be conducted.

For correlation analyses, Pearson's correlation coefficient will be used for normally distributed variables and Spearman's rho for non-normal distributions. The primary analytic focus will be the correlation between LS CE-Chirp ABR amplitudes, latencies, and V/I amplitude ratios and the HINT critical signal-to-noise ratio (SNR-50). Secondary analyses will replicate these correlations for click-evoked ABR parameters. Exploratory analyses will evaluate Wave I amplitude growth functions (µV/dB) and I/V ratio changes across stimulus levels to assess their potential as physiological markers of cochlear synaptopathy.

Effect sizes (Cohen's r or partial η²) and 95 % confidence intervals will accompany all key results. The alpha level will be set at 0.05. Outliers beyond ± 3 SD will be verified and, if necessary, analyzed using robust estimators. Correlation strength will be interpreted according to Cohen's conventions (0.1 = small, 0.3 = medium, 0.5 = large).

Ethical Considerations and Data Handling

All procedures conform to the principles of the Declaration of Helsinki and national ethical guidelines for non-interventional clinical research. Participation is voluntary, and written informed consent will be obtained prior to data collection. Each participant will be assigned a unique numeric code; identifiable information will be stored separately from research data and accessible only to the principal investigator. Data will be encrypted and stored on password-protected institutional drives. Participants may withdraw at any time without penalty. Adverse events or significant discomfort are not anticipated, as ABR and HINT are non-invasive audiological assessments with minimal risk.

Quality Control and Reliability

To ensure data integrity, ABR recordings will be checked for reproducibility by collecting two independent averages per condition. Recordings with residual noise greater than 20 nV or poor inter-replicate correlation (ICC < 0.80) will be excluded. Wave identification will be performed by two trained examiners blinded to group status. Inter-rater reliability for amplitude and latency marking will be calculated. All HINT procedures will follow standardized instructions with the same ambient conditions and calibrated equipment throughout the study.

Expected Outcomes and Significance

The study is expected to demonstrate measurable associations between suprathreshold auditory brainstem response metrics and behavioral speech-in-noise performance. Individuals with suspected hidden hearing loss-particularly those in the speech-in-noise complaint group-are hypothesized to exhibit reduced Wave I amplitudes, lower I/V ratios, and flatter amplitude-growth slopes compared with control participants. These physiological features are predicted to correlate with poorer HINT performance (higher SNR-50 values).

Confirmation of these hypotheses would support the use of LS CE-Chirp ABR as a non-invasive objective tool for identifying neural encoding deficits underlying HHL. The integration of electrophysiological and behavioral outcomes could refine diagnostic criteria for patients who report "I can hear but not understand," despite normal audiograms. Additionally, results may inform future intervention trials aimed at improving neural synchrony or auditory training protocols for individuals with subclinical hearing difficulties.

Study Limitations

The cross-sectional observational design precludes causal inference; however, it is appropriate for hypothesis generation and establishing physiological-behavioral associations. The absence of otoacoustic emission measurements is a potential limitation, but middle-ear status, TEN testing, and normal audiometric thresholds minimize the likelihood of undetected outer-hair-cell dysfunction. Participant numbers are based on power calculations for medium effect sizes; replication with larger cohorts is recommended.

Dissemination Plan

Study findings will be presented at audiology and neuroscience conferences and submitted to peer-reviewed journals indexed in the Science Citation Index Expanded (SCIE). De-identified datasets may be shared upon reasonable request following publication, in accordance with institutional data-sharing policies.

Conclusion

This observational, recruiting study explores how LS CE-Chirp- and Click-evoked ABR parameters relate to speech-in-noise understanding in individuals with suspected hidden hearing loss. By combining objective neural response metrics with subjective and behavioral assessments, the research aims to bridge the gap between physiological evidence of cochlear synaptopathy and functional listening complaints. The expected outcome is an improved framework for early detection of HHL and more precise differentiation of peripheral versus central contributions to speech-in-noise deficits.

ELIGIBILITY:
Inclusion Criteria (Control group):

* Being between 20 and 60 years of age,
* Having bilateral pure-tone audiometry averages (500-1000-2000-4000 Hz) within the normal range (≤25 dB HL),
* Having no tinnitus or auditory complaints,
* Scoring 21 or above on the MoCA test,
* Having no emotional or neurological problems that could interfere with the tests.

Exclusion Criteria (Control group):

* Presence of peripheral and/or central hearing loss,
* Presence of somatosensory tinnitus,
* Presence of emotional and/or neurological problems that could interfere with the tests.

Inclusion Criteria (First study group):

* Being between 20 and 60 years of age,
* Having bilateral pure-tone audiometry averages (500-1000-2000-4000 Hz) within the normal range (≤25 dB HL),
* Having a chronic tinnitus complaint (≥3 months),
* Scoring 21 or above on the MoCA test,
* Having no emotional or neurological problems that could interfere with the tests.

Exclusion Criteria (First study group):

* Presence of peripheral and/or central hearing loss,
* Presence of somatosensory tinnitus,
* Presence of emotional and/or neurological problems that could interfere with the tests.

Inclusion Criteria (Second study group):

* Being between 20 and 60 years of age,
* Having bilateral pure-tone audiometry averages (500-1000-2000-4000 Hz) within the normal range (≤25 dB HL),
* Having no chronic tinnitus complaint,
* Having an average score below 4.3 on the "Speech Perception" subscale of the Speech, Spatial and Qualities of Hearing Scale (SSQ),
* Scoring 21 or above on the MoCA test,
* Having no emotional or neurological problems that could interfere with the tests.

Exclusion Criteria (Second study group):

* Presence of peripheral and/or central hearing loss,
* Presence of somatosensory tinnitus,
* Presence of emotional and/or neurological problems that could interfere with the tests.

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Probability sample method will be used.
Sampling Method: Probability Sample
Enrollment: 63 (Estimated)
Dates: Start 2025-08-20 (Actual); Primary Completion 2026-05-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Correlation between LS CE-Chirp Auditory Brainstem Response (ABR) parameters and Hearing In Noise Test (HINT) performance | Within one month after the completion of participant recruitment.
  This primary outcome will assess the correlation between amplitude (µV) values of Waves I, III, and V, and the V/I amplitude ratio, obtained using LS CE-Chirp-stimulated Auditory Brainstem Response (ABR) at 80, 90, and 100 dB nHL, and the critical signal-to-noise ratio (SNR, dB) obtained from the Hearing In Noise Test (HINT), which evaluates speech understanding in noise.
  ABR recordings will be collected using the Neurosoft Neuro-MEP-4 device, and HINT will be administered in a free-field condition. The degree and direction of correlation between the electrophysiological (ABR) and behavioral (HINT) measures will be analyzed using Pearson or Spearman correlation coefficients, depending on the distribution of the data.

SECONDARY OUTCOMES:
Changes in Wave I amplitude growth and I/V amplitude ratio across stimulus levels in LS CE-Chirp- and Click-evoked ABR | Within one month after completion of participant recruitment.
  This exploratory outcome will examine how Wave I amplitude growth (slope, µV/dB) and I/V amplitude ratio vary across stimulus intensities (80, 90, and 100 dB nHL) in both LS CE-Chirp- and Click-evoked Auditory Brainstem Responses (ABR). These metrics are considered indirect electrophysiological indicators of cochlear synaptopathy or low-spontaneous-rate auditory nerve fiber dysfunction.
  Amplitude values will be measured in microvolts (µV), and stimulus level increments will be expressed in decibels normalized hearing level (dB nHL).
  Analyses will include within-group comparisons of amplitude growth slopes and correlation of these electrophysiological measures with HINT critical SNR (dB) to explore the relationship between suprathreshold neural encoding and speech-in-noise performance.

OTHER OUTCOMES:
Correlation between Click-evoked Auditory Brainstem Response (ABR) parameters and Hearing In Noise Test (HINT) performance | Within one month after completion of participant recruitment.
  This secondary outcome will evaluate the correlation between amplitude (µV) values of Waves I, III, and V, and the V/I amplitude ratio, obtained using Click-evoked Auditory Brainstem Response (ABR) at 80, 90, and 100 dB nHL, and the critical signal-to-noise ratio (SNR, dB) obtained from the Hearing In Noise Test (HINT), which assesses speech understanding in noise.
  ABR measurements will be recorded using the Neurosoft Neuro-MEP-4 device, and HINT will be conducted in a free-field setup. The degree and direction of correlation between electrophysiological (ABR) and behavioral (HINT) measures will be analyzed using Pearson or Spearman correlation coefficients, depending on data normality.

CONTACTS AND LOCATIONS:
Overall Officials: Eyyup Kara, Asst. Prof., Study Chair — Istanbul University - Cerrahpasa
Locations (1):
- Istanbul University-Cerrahpaşa, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Kara E, Aydin K, Akbulut AA, Karakol SN, Durmaz S, Yener HM, Gozen ED, Kara H. Assessment of Hidden Hearing Loss in Normal Hearing Individuals with and Without Tinnitus. J Int Adv Otol. 2020 Apr;16(1):87-92. doi: 10.5152/iao.2020.7062. PMID 32209515
- [Result] Lobarinas E, Salvi R, Ding D. Selective Inner Hair Cell Dysfunction in Chinchillas Impairs Hearing-in-Noise in the Absence of Outer Hair Cell Loss. J Assoc Res Otolaryngol. 2016 Apr;17(2):89-101. doi: 10.1007/s10162-015-0550-8. Epub 2015 Dec 21. PMID 26691159
- [Result] Kujawa SG, Liberman MC. Adding insult to injury: cochlear nerve degeneration after "temporary" noise-induced hearing loss. J Neurosci. 2009 Nov 11;29(45):14077-85. doi: 10.1523/JNEUROSCI.2845-09.2009. PMID 19906956
- [Result] Chambers AR, Resnik J, Yuan Y, Whitton JP, Edge AS, Liberman MC, Polley DB. Central Gain Restores Auditory Processing following Near-Complete Cochlear Denervation. Neuron. 2016 Feb 17;89(4):867-79. doi: 10.1016/j.neuron.2015.12.041. Epub 2016 Jan 28. PMID 26833137
- [Result] Gratias P, Nasr J, Affortit C, Ceccato JC, Francois F, Casas F, Pujol R, Pucheu S, Puel JL, Wang J. Impulse Noise Induced Hidden Hearing Loss, Hair Cell Ciliary Changes and Oxidative Stress in Mice. Antioxidants (Basel). 2021 Nov 25;10(12):1880. doi: 10.3390/antiox10121880. PMID 34942983
- [Result] Lopez-Poveda EA. Why do I hear but not understand? Stochastic undersampling as a model of degraded neural encoding of speech. Front Neurosci. 2014 Oct 30;8:348. doi: 10.3389/fnins.2014.00348. eCollection 2014. PMID 25400543
- [Result] Liu J, Stohl J, Overath T. Hidden hearing loss: Fifteen years at a glance. Hear Res. 2024 Mar 1;443:108967. doi: 10.1016/j.heares.2024.108967. Epub 2024 Jan 30. PMID 38335624